CLINICAL TRIAL: NCT07201675
Title: Vedisertib (RC48/ADC) Combined With Toripalimab in Bladder-preserving Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSZ05
Record Dates: First submitted 2025-09-07; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Muscle Invasive Bladder Cancer (MIBC)
Keywords: RC48; muscle invasive bladder cancer; Toripalimab
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC combined with toripalimab for bladder-sparing therapy (Experimental)
  Interventions: Drug: RC48-ADC combined with toripalimab for bladder-sparing therapy

INTERVENTIONS:
Drug: RC48-ADC combined with toripalimab for bladder-sparing therapy — RC48-ADC combined with toripalimab for bladder-sparing therapy

SUMMARY:
This is a phase II clinical study to evaluate the efficacy of RC48-ADC combined with toripalimab bladder-sparing therapy.

The RC48-ADC dose in this study is 2.0 mg/kg Q2W and toripalimab is 3 mg/kg Q2W.

This study plans to enroll 59 participants. The participants will start drug therapy within 2 weeks after the first diagnostic resection in the first stage, receiving RC48-ADC combined with toripalimab 3 times. At the 8th week after enrollment, the second stage of cystectomy was performed, and RC48-ADC combined with toripalimab was treated every two weeks thereafter for a total of 3 treatments. After the completion of the two-stage treatment, the participants should be discharged from the group by cystoscopy or other imaging examinations. On the contrary, if the participants have complete remission or partial remission, continue to the third stage of treatment, that is, receive RC48-ADC combined with toripalimab every two weeks for a total of 6 treatments, followed by cystoscopy, imaging, or a third cystectomy. If the participants achieve complete remission of the disease, maintenance immunotherapy will be given for 12 months. If the participants show that there is still a tumor, the participants will be discharged from the group for other treatments. Due to disease progression, death, participants voluntarily requested termination of study treatment, toxicity intolerance, initiation of new anti-tumor therapy, pregnancy, serious violation of the study process stipulated by the protocol, termination of study treatment determined by the investigator based on the best interests of the participants, loss to follow-up, whichever occurred first.

During the study, the first and second electrotoxic tissues were sequenced using RNA and single-cell sequencing, and ctDNA was tested in urine before treatment, in the third month, and in the sixth month.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign the informed consent form;
2. Male or female, age ≥ 18 years;
3. Expected survival ≥ 18 months;
4. Pathological and imaging diagnosis of cT2-4aN0M0MIBC;
5. Subjects are able to provide specimens of tumor primary lesions detected by PD-L1 and HER2; HER2 IHC 1 or 2 or 3 ;
6. No previous systemic therapy;
7. ECOG performance status score of 0 or 1 point;
8. Adequate cardiac, bone marrow, liver, and renal function (based on normal values at the study center):

   1. Left ventricular ejection fraction ≥50%;
   2. Hemoglobin ≥9 g/dL;
   3. Absolute neutrophil count (ANC) ≥ 1.5×109/L;
   4. Platelets≥ 100 ×109/L;
   5. In patients without liver metastasis, serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN); Blood in liver metastases
   6. Clear total bilirubin ≤3× ULN
   7. ALT and AST ≤2.5 × ULN in the absence of liver metastases, ALT and AST≤5 × ULN in the presence of liver metastases;
   8. Serum creatinine ≤1.5× ULN;
9. For female subjects: should be zsurgically sterile, postmenopausal patients, or agree to use at least one medically approved contraceptive measure (such as intrauterine device [IUD], birth control pills, or condoms) during the study treatment period and for 6 months after the end of the study treatment period, must have a negative serum or urine pregnancy test within 7 days prior to study enrollment, and must be non-lactating. Male subjects should agree to use at least one medically approved contraceptive measure (such as condoms, abstinence, etc.) during the study treatment period and within 6 months after the end of the study treatment period;
10. Willing and able to comply with trial and follow-up procedures.

Exclusion Criteria:

1. History of malignant tumors other than urothelial carcinoma, except for the following two conditions:

   1. Patients have received potentially curative therapy and no evidence of the disease within 5 years;
   2. Successfully undergoing resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, and other carcinomas in situ;
2. Suffering from diseases that affect the absorption, distribution, metabolism or clearance of the study drug (such as severe vomiting, chronic diarrhea, intestinal obstruction, malabsorption, etc.);
3. Previous allogeneic stem cell or parenchymal organ transplantation; Patients who have received other anti-tumor systemic therapy (including traditional Chinese medicine with anti-tumor indications) in the past, less than 4 weeks after the completion of treatment to before the use of this study, or who have not recovered to ≤ CTCAE grade 1 (except for alopecia and pigmentation);
4. Previous or current congenital or acquired immunodeficiency disease;
5. Active or previous documented autoimmune or inflammatory diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, hypophysitis, hyperthyroidism or hypothyroidism, asthma requiring bronchodilator treatment, etc.), vitiligo or asthma that has been completely resolved in childhood, and those who do not need any intervention in adulthood can be included;
6. Use of systemic immunosuppressive drugs within 2 weeks prior to enrollment, or anticipation of need for systemic immunosuppressive drugs during the study, except for the following:

   1. intranasal, inhaled, topical, or local injections (such as intra-articular injections) corticosteroids;
   2. Systemic corticosteroids at doses not exceeding 10 mg/day of prednisone or other equivalent effects;
   3. prophylactic use of corticosteroids for hypersensitivity;
7. Patients have a known or suspected history of allergy to vidicitumab, anti-PD-1 drugs, or a history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or allergic to the excipients of the study drug;
8. Thrombotic or thromboembolic events within the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc.;
9. Patients at risk of severe bleeding evaluated by doctors, including but not limited to severe bleeding (bleeding within 3 months> 30 ml), hemoptysis (bleeding within 4 weeks> 5 ml), if the above conditions occur, gastroscopy/evaluation can be performed, and the microscopic evaluation shall prevail; or have active bleeding or abnormal coagulation function, have a bleeding tendency or are receiving thrombolytic, anticoagulant or antiplatelet therapy;
10. Significant clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina or coronary artery bypass grafting within the past 6 months, congestive heart failure (NYHA classification> of the New York Heart Association Grade 2), poorly controlled or arrhythmias requiring pacemaker therapy, hypertension that cannot be controlled by medication (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg);
11. Other significant clinical and laboratory abnormalities that the investigator believes to affect the safety evaluation, such as: uncontrollable diabetes, chronic kidney disease, grade II or above peripheral neuropathy (CTCAE V5.0), abnormal thyroid function, etc.;
12. Serious infection in the active phase or poorly controlled clinically; Active infection, including:

    1. HIV (HIV) (HIV1/2 antibody) positive;
    2. Active hepatitis B (HBsAg positive or HBV DNA>2000IU/ml with abnormal liver function);
    3. Active hepatitis C (positive HCV antibody or HCV RNA ≥103 copies/ml with abnormal liver function);
    4. Active tuberculosis;
    5. Other uncontrollable active infections (CTCAE V5.0 >2);
13. Not yet recovered from surgery, such as unhealed incisions or serious postoperative complications;
14. Pregnant or lactating women, as well as female or male patients of childbearing potential who are unwilling or unable to take effective contraceptive measures;
15. Other conditions that the investigator deems unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
cCR (Clinical Complete response) | From date of randomization, follow-up once every 12 weeks until the date of first documented death, loss to follow-up, withdrawal of informed consent, whichever came first, assessed up to 60 months

SECONDARY OUTCOMES:
OS (Overall Survival) | From date of randomization, follow-up once every 12 weeks until the date of first documented death, loss to follow-up, withdrawal of informed consent, whichever came first, assessed up to 60 months
DFS (Disease Free Survival) | From date of randomization, follow-up once every 12 weeks until the date of first documented death, loss to follow-up, withdrawal of informed consent, whichever came first, assessed up to 60 months
cPR (Clinical Partial Response) | From date of randomization, follow-up once every 12 weeks until the date of first documented death, loss to follow-up, withdrawal of informed consent, whichever came first, assessed up to 60 months
Barthel Index | From date of randomization, follow-up once every 12 weeks until the date of first documented death, loss to follow-up, withdrawal of informed consent, whichever came first, assessed up to 60 months
  BI (Barthel Index), 0-100 score. The higher the score, the stronger the ability to take care of oneself.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sheng X, Wang L, He Z, Shi Y, Luo H, Han W, Yao X, Shi B, Liu J, Hu C, Liu Z, Guo H, Yu G, Ji Z, Ying J, Ling Y, Yu S, Hu Y, Guo J, Fang J, Zhou A, Guo J. Efficacy and Safety of Disitamab Vedotin in Patients With Human Epidermal Growth Factor Receptor 2-Positive Locally Advanced or Metastatic Urothelial Carcinoma: A Combined Analysis of Two Phase II Clinical Trials. J Clin Oncol. 2024 Apr 20;42(12):1391-1402. doi: 10.1200/JCO.22.02912. Epub 2023 Nov 21. PMID 37988648
- [Background] Wang J, Liu Y, Zhang Q, Li W, Feng J, Wang X, Fang J, Han Y, Xu B. Disitamab vedotin, a HER2-directed antibody-drug conjugate, in patients with HER2-overexpression and HER2-low advanced breast cancer: a phase I/Ib study. Cancer Commun (Lond). 2024 Jul;44(7):833-851. doi: 10.1002/cac2.12577. Epub 2024 Jun 28. PMID 38940019
- [Background] Sheng X, Chen H, Hu B, Yao X, Liu Z, Yao X, Guo H, Hu Y, Ji Z, Luo H, Shi B, Liu J, Wu J, Zhou F, He Z, Fan J, Wang W, Feng H, Yao S, Keegan P, Huang Y, Guo J. Safety, Efficacy, and Biomarker Analysis of Toripalimab in Patients with Previously Treated Advanced Urothelial Carcinoma: Results from a Multicenter Phase II Trial POLARIS-03. Clin Cancer Res. 2022 Feb 1;28(3):489-497. doi: 10.1158/1078-0432.CCR-21-2210. Epub 2021 Nov 5. PMID 34740921